CLINICAL TRIAL: NCT03623308
Title: Microbiome Stability After Addition of a High Fiber, Whole Grain and Bran Cereal to the Diets of Healthy Individuals
Brief Title: Whole Grain and Fiber Addition Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: General Mills (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00002230
Record Dates: First submitted 2018-04-12; First posted 2018-08-09 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiber Intervention I (Experimental): Participants will be asked to consume two ½ cup servings of fiber cereal daily (equivalent to 28 g fiber) for 14 days, one in the morning and one in the evening.
  Interventions: Other: Fiber cereal
- Fiber Intervention II (Experimental): Participants will be asked to consume two ¼ cup servings of fiber cereal daily (equivalent to 14 g fiber) for 14 days, one in the morning and one in the evening.
  Interventions: Other: Fiber cereal

INTERVENTIONS:
Other: Fiber cereal — Whole grain and bran cereal

SUMMARY:
The human gut microbiota is the complex community of bacteria that reside within the human gastrointestinal tract. This community plays an important role in supporting normal immune function and digestion. Disruption of the microbial communities within the gastrointestinal tract, sometimes termed "dysbiosis" is linked to a wide range of human diseases, including obesity, metabolic syndrome, malnutrition, and cancer. Stability of the microbiome is thought to be important for human health, however the factors that drive microbiome community stability are poorly understood.

Within the gastrointestinal tract, the microbiota is constantly exposed to complex mixtures of foods and the products of digestion. Importantly, changes in diet have been shown to rapidly induce shifts in microbial community composition. These compositional shifts can also affect microbial production of bioactive metabolites, which may be one mechanism to explain how the microbiome impacts host physiology and disease.

Fiber is often considered to be one of the largest contributors to microbial compositional shifts that follow dietary interventions. Fiber resists digestion and persists through the gastrointestinal tract to reach the large intestine where it can be metabolized by bacteria. The end products of this metabolism are the short chain fatty acids (SCFAs), acetate and butyrate, which are often associated with beneficial health outcomes. Fibrous foods are also a source of polyphenols and other phenolic compounds that may be used by microbes in the production of secondary metabolites or freed from the food matrix by microbial enzymes.

The purpose of this study is to: 1) to investigate the impact of high fiber, whole grain and bran cereal on microbiome stability, and 2) to explore the microbial contribution to polyphenol metabolism from whole grain in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults over 18 years
* BMI between 18 and 30
* English speaker with ability to use a computer/smartphone.

Exclusion Criteria:

* Women who are currently pregnant or breastfeeding
* Current use of antibiotics or use of antibiotics within the last month
* Self-reported, pre-existing history of gastrointestinal disease including IBD, IBS, Crohn's disease, Celiac disease (or self-reported sensitivity to gluten), history of bowel blockage/impacted stool, fecal incontinence, gastroparesis or diverticulosis.
* Type I/II diabetes mellitus
* Participants actively trying to lose weight
* Chronic use of antacids and/or laxatives
* Use of seizure disorder medications or tricyclic antidepressants
* Consumption of drugs or supplements related to energy intake (i.e. diet pills and appetite suppressants)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Change in microbiome stability | Change from baseline to 6 weeks
  Shotgun metagenomic sequencing of stool samples

SECONDARY OUTCOMES:
Microbiome functional capacity | Baseline, 2 weeks, 6 weeks
  Assessment of microbiome functional capacity using DNA alignment to KEGG orthology
Urinary metabolome | Baseline, 2 weeks, 6 weeks
  Targeted liquid chromatography mass spectroscopy to detect urinary metabolites
Fecal short chain fatty acids | Baseline, 2 weeks, 6 weeks
  Targeted liquid chromatography mass spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code